CLINICAL TRIAL: NCT01396252
Title: Randomized, Placebo-Controlled, Double-Blind, Ascending Multiple-Dose Study to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamics of BMS-820836 in Healthy Japanese Subjects and Japanese Patients With Depression
Brief Title: Japanese Phase 1 Multiple Ascending Dose (MAD) Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CN162-014
Record Dates: First submitted 2011-07-15; First posted 2011-07-18 (Estimated); Last update posted 2013-06-10 (Estimated); Status verified 2013-06

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — 6-(2-methyl-4-(2-naphthyl)-1,2,3,4-tetrahydroisoquinolin-7-yl)pyridazin-3-amine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm1: BMS-820836 (Experimental): Panels 1-4 are fixed dose panels (0.5, 1, 1 and 2 mg respectively), Panels 5-7 are titration dose panels (initiated at 1 mg and dose escalated to the target dose of 2 mg)
  Interventions: Drug: BMS-820836
- Arm 2: Placebo matching BMS-820836 (Placebo Comparator): Panels 1-4 are fixed dose panels (0.5, 1, 1 and 2 mg respectively), Panels 5-7 are titration dose panels (initiated at 1 mg and dose escalated to the target dose of 2 mg)
  Interventions: Drug: Placebo matching BMS-820836

INTERVENTIONS:
Drug: BMS-820836 — Tablets, Oral, 0.5 mg, Once daily, 14 days
  Arms: Arm1: BMS-820836
Drug: BMS-820836 — Tablets, Oral, 1 mg, Once daily, 14 days
  Arms: Arm1: BMS-820836
Drug: BMS-820836 — Tablets, Oral, 2 mg, Once daily, 14 days
  Arms: Arm1: BMS-820836
Drug: Placebo matching BMS-820836 — Tablets, Oral, 0 mg, Once daily, 14 days
  Arms: Arm 2: Placebo matching BMS-820836
Drug: BMS-820836 — Tablets, Oral, (initiated at 1 mg and dose escalated to the target dose of 2 mg), Once daily, 14 days
  Arms: Arm1: BMS-820836

SUMMARY:
The purpose of this clinical study is to assess the safety and tolerability of multiple oral doses of BMS-820836 in healthy Japanese subjects and Japanese patients with depression.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Japanese subjects and Japanese patients with depression (Hamilton Rating Scale for Depression (HAM-D) ≥ 14), ages 20 to 55 years.

Exclusion Criteria:

* Any significant acute or chronic medical illness.
* Non-compliance, or overall not suitable as determined by the investigator.
* History of, or current clinically significant psychiatric disorders or illnesses, substance abuse or dependence.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2011-09; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability based on medical review of adverse events & results of vital sign measurements, electrocardiogram (ECGs), physical examinations, clinical laboratory test, suicidality evaluation & Montgomery Asberg Depression Rating Scale (MADRS) | Day 1 through Day 33

SECONDARY OUTCOMES:
Multiple-dose pharmacokinetics parameter Maximum observed concentration (Cmax) of BMS-820836 and BMS-821007 | Day1 through Day 33
Multiple-dose pharmacokinetics parameter Concentration at 24 h (C24) of BMS-820836 and BMS-821007 | Day1 through Day 33
Multiple-dose pharmacokinetics parameter Time of maximum observed concentration (Tmax) of BMS-820836 and BMS-821007 | Day1 through Day 33
Multiple-dose pharmacokinetics parameter Area under the concentration-time curve in one dosing interval (AUC(TAU)) of BMS-820836 and BMS-821007 | Day1 through Day 33
Multiple-dose pharmacokinetics parameter Apparent total body clearance (CLT/F) of BMS-820836 and BMS-821007 | Day1 through Day 33
Multiple-dose pharmacokinetics parameter accumulation index (AI) of BMS-820836 and BMS-821007 | Day1 through Day 33
Multiple-dose pharmacokinetics parameter half-life (T-HALF) of BMS-820836 and BMS-821007 | Day1 through Day 33
Multiple-dose pharmacokinetics parameter Molar ratio of metabolite to parent Cmax or AUC(TAU) | Day1 through Day 33
ECG parameters (heart rate, PR, QRS, QT, and QTcF intervals) | Day1 through Day 33
  QTcF intervals - QT interval corrected for heart rate according to Fridericia's formula
Vital sign measures (heart rate and blood pressure) and the orthostatic changes | Day1 through Day 33

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Taito-Ku, Tokyo, Japan

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx